CLINICAL TRIAL: NCT05612035
Title: A Phase 2a Randomized, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of MK-5475 in Adults With Pulmonary Hypertension Associated With Chronic Obstructive Pulmonary Disease
Brief Title: Frespaciguat (MK-5475) INSIGNIA-PH-COPD: A Study of the Efficacy and Safety of Frespaciguat (an Inhaled sGC Stimulator) in Adults With PH-COPD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5475-013; MK-5475-013 (Other: MSD); 2022-501201-13-00 (Registry Identifier: EU CT); U1111-1279-8512 (Registry Identifier: UTN)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frespaciguat (Experimental): Participants with PH-COPD will receive 380 µg of frespaciguat as an oral inhalation once daily for 24 weeks (base period) and thereafter for up to 42 months (optional extension period).
  Interventions: Drug: Frespaciguat
- Placebo (Placebo Comparator): Participants with PH-COPD will receive matching placebo as an oral inhalation once daily for 24 weeks (base period) and then 380 µg of frespaciguat as an oral inhalation once daily for up to 42 months (optional extension period).
  Interventions: Drug: Frespaciguat; Drug: Placebo

INTERVENTIONS:
Drug: Frespaciguat — Frespaciguat 380 µg administered as dry powder inhalation once daily.
  Other Names: MK-5475
Drug: Placebo — Placebo administered as dry powder inhalation once daily.
  Arms: Placebo

SUMMARY:
Researchers are looking for ways to treat pulmonary hypertension (PH) caused by chronic obstructive pulmonary disease (COPD). The goal of the study is to learn if people who take frespaciguat can walk farther in 6 minutes at Week 24 compared to people who take placebo.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has Group 3.1 pulmonary hypertension chronic obstructive pulmonary disease (PH-COPD) as defined by the Clinical Classification of Pulmonary Hypertension.
* Has a right heart catheterization (RHC) at screening or historical RHC within 12 months before screening that meets hemodynamic criteria.
* Has a physician diagnosis of obstructive lung disease on pulmonary function testing (PFT) performed at screening.
* Has a WHO Functional Class assessment of Class II to IV.
* If on supplemental oxygen, the regimen must be stable.
* Has stable and optimized chronic, baseline COPD-specific therapy.
* If on PDE5 inhibitor, has stable concomitant use (initiated at least 3 months prior to randomization and no change in drug or dosage for at least 3 months prior to randomization) and changes to PDE5 inhibitor dosing is not anticipated during the 24 week Base Period.
* If on antihypertensives and/or a diuretic regimen has stable concomitant use.
* If on anticoagulants has stable concomitant use.
* Is of any sex/gender from 40 to 85 years of age inclusive.
* Female is not pregnant or breastfeeding, and is not of childbearing potential or uses acceptable contraceptive method or abstains from sexual intercourse, or has a negative highly sensitive pregnancy test within 24 hours before the first dose of study intervention, or whose history and sexual activity has been reviewed by the investigator.

Exclusion criteria:

* Has Group 1 pulmonary arterial hypertension (PAH), Groups 2, 4 or 5 pulmonary hypertension (PH).
* Has non-COPD related Group 3 PH.
* Has evidence of untreated more than mild obstructive sleep apnea.
* Has significant left heart disease.
* Expects to receive a lung and/or heart transplant from screening through the end of the 24 week Base Period.
* Has evidence of a resting oxygen saturation (SpO2) < 88%.
* Has experienced a moderate or severe COPD exacerbation within 2 months before randomization.
* Has experienced right heart failure within 2 months before randomization.
* Has uncontrolled tachyarrhythmia.
* Has acute coronary syndrome, undergone coronary artery bypass graft, or percutaneous coronary intervention within 2 months before randomization.
* Has evidence of significant chronic renal insufficiency.
* Has evidence of chronic liver disease, portal hypertension, cirrhosis, or hepatic abnormalities.
* Initiated a pulmonary rehabilitation program within 2 months before randomization.
* Has impairments that limit the ability to perform 6MWT.
* Has history of cancer.
* Is a user of illicit drugs or has a recent history of drug/alcohol abuse or dependence.
* Has used PAH-specific therapies within 2 months of randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2029-10-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in 6-minute Walk Distance (6MWD) at Week 24 | Baseline and Week 24
  6MWD is assessed using the 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Mean Change From Baseline in 6MWD at Week 12 | Baseline and Week 12
  6MWD is assessed using the 6-minute walk test (6MWT).
Mean Change From Baseline in N-Terminal Pro B-Type Natriuretic Peptide (NT-proBNP) at Week 12 | Baseline and Week 12
  NT-proBNP was measured at baseline and Week 12.
Mean Change From Baseline in NT-ProBNP at Week 24 | Baseline and Week 24
  NT-proBNP was measured at baseline and Week 24
Percentage of Participants Whose World Health Organization-Functional Class (WHO-FC) Does not Worsen Relative to Baseline at Week 12 | Baseline and Week 12
  Participants are assigned one of four WHO-FC, dependent on limits of physical activity. As WHO-FC increases from I to IV, limits of physical activity increase.
Percentage of Participants Whose WHO-FC Does not Worsen Relative to Baseline at Week 24 | Baseline and Week 24
  Participants are assigned one of four WHO-FC, dependent on limits of physical activity. As WHO-FC increases from I to IV, limits of physical activity increase.
Percentage of Participants With One or More Adverse Events (AEs) | Up to Week 206
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Percentage of Participants who Discontinued Study Treatment due to an AE | Up to Week 204
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (84):
- United States (18):
  - UCSF Helen Diller Medical Center at Parnassus Heights ( Site 0110), San Francisco, California
  - University of Colorado Anschutz Medical Campus-University of Colorado Hospital Cardiac and Vascular ( Site 0101), Aurora, Colorado
  - Clinovation Intl. Corp. ( Site 0108), Sebring, Florida
  - Alexian Brothers Medical Center-Pulmonary ( Site 0109), Elk Grove Village, Illinois
  - University of Iowa ( Site 0103), Iowa City, Iowa
  - University of Kansas Medical Center-IM-Pulmonary and Critical Care Medicine ( Site 0102), Kansas City, Kansas
  - Lexington VA Medical Center - Cooper Division ( Site 0137), Lexington, Kentucky
  - Corewell Health ( Site 0133), Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Minnesota ( Site 0131), Rochester, Minnesota
  - Creighton University Clinical Research Office ( Site 0123), Omaha, Nebraska
  - University of New Mexico Hospital ( Site 0146), Albuquerque, New Mexico
  - UNC Health - Eastowne Medical Office-Clinical Trials Unit ( Site 0147), Chapel Hill, North Carolina
  - Temple University Hospital ( Site 0104), Philadelphia, Pennsylvania
  - UPMC Montefiore University Hospital-Department of Medicine ( Site 0149), Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center ( Site 0114), Dallas, Texas
  - The University of Texas Health Science Center at Houston ( Site 0105), Houston, Texas
  - Intermountain Medical Center-Division of Pulmonary & Critical Care Medicine ( Site 0140), Murray, Utah
  - University of Virginia Health System-Division of Pulmonary and Critical Care Medicine ( Site 0111), Charlottesville, Virginia
- Argentina (5):
  - Fundación Respirar ( Site 0305), CABA, Buenos Aires
  - Centro Medico Capital ( Site 0301), La Plata, Buenos Aires
  - Instituto de Cardiologia de Tucuman-Area de Investigacion Clinica ( Site 0303), San Miguel de Tucumán, Tucumán Province
  - Hospital Britanico de Buenos Aires ( Site 0307), CABA
  - Hospital Privado Universitario de Córdoba-Clinical Cardiology Department ( Site 0302), Córdoba
- Australia (5):
  - Royal Prince Alfred Hospital-Department of Respiratory Medicine ( Site 0903), Camperdown, New South Wales
  - Westmead Hospital ( Site 0902), Westmead, New South Wales
  - WESLEY RESEARCH INSTITUTE Limited ( Site 0906), Auchenflower, Queensland
  - The Prince Charles Hospital ( Site 0904), Brisbane, Queensland
  - Mater Misericordiae Limited ( Site 0905), South Brisbane, Queensland
- Austria (2):
  - Medizinische Universität Graz-Klinische Abteilung für Pulmonologie ( Site 1201), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 1202), Innsbruck, Tyrol
- Belgium (2):
  - Université Libre de Bruxelles - Hôpital Erasme ( Site 1302), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven ( Site 1301), Leuven, Vlaams-Brabant
- Colombia (4):
  - Clinica Cardio VID ( Site 0504), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0508), Barranquilla, Atlántico
  - Fundación Valle del Lili ( Site 0509), Cali, Valle del Cauca Department
  - Centro de Investigaciones Clinicas SAS ( Site 0505), Cali, Valle del Cauca Department
- France (5):
  - C.H.U Hôpital Nord ( Site 1503), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois ( Site 1502), Vandœuvre-lès-Nancy, Lorraine
  - CHU Angers ( Site 1506), Angers, Maine-et-Loire
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre-Pneumologie ( Site 1501), Le Kremlin-Bicêtre, Paris
  - Centre Hospitalier Universitaire de Poitiers ( Site 1505), Poitiers, Vienne
- Germany (5):
  - Thoraxklinik-Heidelberg gGmbH-Zentrum für Pulmonale Hypertonie ( Site 1603), Heidelberg, Baden-Wurttemberg
  - UKGM Gießen/Marburg ( Site 1604), Giessen, Hesse
  - Medizinische Hochschule Hannover ( Site 1602), Hanover, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden ( Site 1601), Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein-Pneumologie ( Site 1605), Lübeck, Schleswig-Holstein
- Guatemala (4):
  - Unidad De Diagnostico Cardiologico-Unidad de Diagnostico Cardiologico ( Site 0605), Guatemala City
  - MEDI-K ( Site 0607), Guatemala City
  - Clinica Medica ( Site 0601), Guatemala City
  - Private Practice - Dr. Jeremias Guerra Mejia ( Site 0603), Guatemala City
- Israel (2):
  - Rambam Health Care Campus ( Site 1701), Haifa
  - Rabin Medical Center ( Site 1702), Petah Tikva
- Italy (3):
  - Cattinara Hospital ( Site 1801), Trieste, Friuli Venezia Giulia
  - Ospedale San Gerardo-ASST Monza-Cardio Vasolare- Clinica pneumologica ( Site 1802), Monza, Lombardy
  - ISMETT Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione ( Site 1804), Palermo
- Mexico (4):
  - Centro Médico Nacional Siglo XXI ( Site 0708), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0704), Mexico City, Mexico City
  - INVECORDIS S.C. ( Site 0703), Hacienda de Las Palmas, State of Mexico
  - Instituto Nacional de Cardiologia Ignacio Chavez ( Site 0701), México
- Peru (3):
  - Unidad de Investigacon de la Clinica Internacional ( Site 0804), Lima Cercado, Lima region
  - Clinica Ricardo Palma-Centro de Investigacion de Enfermedades Respiratorias Thorax ( Site 0806), San Isidro, Lima region
  - Clínica Providencia ( Site 0803), San Miguel, Lima region
- South Africa (4):
  - Charlotte Maxeke Johannesburg Academic Hospital ( Site 2108), Johannesburg, Gauteng
  - Netcare Milpark Hospital ( Site 2103), Johannesburg, Gauteng
  - Netcare St Augustine's Hospital ( Site 2105), Durban, KwaZulu-Natal
  - TREAD Research ( Site 2101), Cape Town, Western Cape
- South Korea (4):
  - Gachon University Gil Medical Center ( Site 1101), Namdong-gu, Incheon
  - Seoul National University Hospital ( Site 1103), Seoul
  - Asan Medical Center ( Site 1102), Seoul
  - Samsung Medical Center ( Site 1104), Seoul
- Spain (5):
  - Hospital Universitario Marqués de Valdecilla-Pneumology ( Site 2003), Santander, Cantabria
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 2001), Barcelona, Catalonia
  - Parc de Salut Mar - Hospital del Mar ( Site 2006), Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 2002), Barcelona
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 2005), Seville
- Switzerland (3):
  - University Hospital Basel ( Site 2205), Basel, Canton of Basel-City
  - UniversitätsSpital Zürich ( Site 2201), Zurich, Canton of Zurich
  - Cantonal Hospital St.Gallen ( Site 2203), Sankt Gallen
- Turkey (Türkiye) (4):
  - Hacettepe Universite Hastaneleri ( Site 2301), Ankara
  - Ankara Bilkent Şehir Hastanesi. ( Site 2307), Ankara
  - Eskisehir Osmangazi University-Cardiology ( Site 2304), Eskişehir
  - Istanbul Universitesi Istanbul Tıp Fakultesi Hastanesi-Chest Disease ( Site 2302), Istanbul
- United Kingdom (2):
  - Hammersmith Hospital-Department of Cardiology ( Site 2401), London, London, City of
  - Sheffield Teaching Hospitals NHS Foundation Trust-Clinical Research Facility ( Site 2405), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26243&tenant=MT_MSD_9011